CLINICAL TRIAL: NCT05260398
Title: Examining the Impacts on In-School Behaviors of In-Home Engagement With a Biofeedback-based Videogame Application
Brief Title: Examining the Impacts on In-School Behaviors of In-Home Videogame Play
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neuromotion Labs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1076MIGH22
Record Dates: First submitted 2022-02-07; First posted 2022-03-02 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Emotional Regulation; Problem Behavior; Irritable Mood
MeSH Terms: conditions — Emotional Regulation; Problem Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Enrolled family random study cohort assignment will be masked from school teachers, who will complete outcome measure questionnaires about enrolled child participants at baseline and follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mightier Now (Experimental): 8 weeks of use ad-libitum. Parents will be encouraged to have their children play Mightier games at least 3 times a week (totalling 45 minutes or more of play each week) for the 8-week duration.
  Interventions: Behavioral: Mightier Online Gameplay
- Mightier Later (No Intervention): 8 weeks of wait list. Families in the Mightier Later condition will receive their Mightier shipment and will be encouraged to play Mightier after follow-up questionnaires have been completed 8 weeks after parents and teachers complete baseline questionnaires.

INTERVENTIONS:
Behavioral: Mightier Online Gameplay — Mightier is a video-game-based biofeedback intervention that capitalizes on children's love of video games to increase emotional awareness and facilitate emotion regulation practice through heart rate (HR) control. Each family receives a Mightier Kit (Mighty Band heart rate monitor, dedicated Mightier tablet unless the family prefers to use their own device) and the Mightier App. Children wear a "Mighty Band" heart rate monitor on their arm while they play any one of 26+ games. As their heart rate rises the games become more difficult. For example, during a cooking game, smoke may appear on the screen and obscure the player's view. Children can either opt into an explicit cool down activity (deep breathing, progressive muscle relaxation, crossing the midline, or visualization) or cool down on their own. By simply playing Mightier, children are motivated to practice calming strategies in moments of challenge.
  Arms: Mightier Now

SUMMARY:
The proposed study aims to investigate the effects of children's in-home engagement with a biofeedback video game-based intervention on children's in-school behaviors. For the proposed study, families with no prior Mightier exposure will engage in online gameplay for eight weeks. Mightier will recruit families through social media and clinical settings, then Mightier will randomly assign participants to one of two groups: a group in which the child participant is encouraged to play Mightier games with biofeedback elements 45 or more minutes a week, broken into 3 or more sessions a week soon after baseline data have been collected, and a group in which the child participant receives Mightier and is invited to play Mightier games with biofeedback elements after all study baseline and follow-up data have been collected. The investigators will aim to enroll 20 parent-child dyads in each group.

Specific Aims and Hypotheses:

1. Demonstrate that child engagement in Mightier biofeedback video games is correlated to child improvement in school behaviors. The investigators hypothesize that teachers of child participants will report reductions in child school behavior challenges after 8 weeks of child Mightier gameplay.
2. Demonstrate that child engagement in Mightier biofeedback video games is correlated to child improvement in at-home behaviors and general improvement in emotion regulation. The investigators hypothesize that parents of child participants will report a reduction in child behavior challenges and improvements in child emotion regulation after 8 weeks of child Mightier gameplay.

DETAILED DESCRIPTION:
Study Design:

A randomized controlled trial comparing pre- and post-measures for a group in which child participants play Mightier video games for the active 8-week study period (Mightier Now group) to a group in which child participants wait during the active 8-week study period, then play Mightier after post-measures are collected (Mightier Later group).

Study Sample:

40 parent-child dyads in which the enrolled children are between 6 and 11 years old, have no prior Mightier experience, and attend school outside the home; 40 school teacher informants, who will complete baseline and follow-up measures on behalf of enrolled children.

Study Aims:

Aim 1. Demonstrate that children's in-home Mightier play is associated with reduced in-school emotional and behavioral problems. The investigators hypothesize that teachers will report reductions in child participants' school emotional and behavioral challenges after 8 weeks of child Mightier gameplay at home.

Aim 2. Demonstrate that children's in-home Mightier play is associated with parent-perceived reductions in child emotional and behavioral challenges and overall improvements in child emotion regulation. The investigators hypothesize that parents will report reductions in child participants' emotional and behavioral challenges and improvements in child emotion regulation after 8 weeks of child Mightier gameplay.

Recruitment Participants will be recruited to the study via social media ads, emails to families who have inquired about Mightier research studies, and clinician and educator referrals.

Screening Families who are interested in enrolling in the study will complete screening via an online questionnaire form to screen for inclusion and exclusion criteria.

During study screening, families will be given a link to share with their child's school teacher, along with sample language that families can use to inform the teacher that the family would like to participate in a research study, that the study requires data at baseline and Week 8 from questionnaires completed by a teacher who sees the student regularly.

Teachers who use the link provided by families who are interested in the study will link to a web page providing information about the research study and asking is the teacher is willing and able to complete study measures.

If children meet inclusion/exclusion criteria and teachers are willing and able to complete questionnaires, then parents/guardians and child participants will be invited to schedule a video call to complete study informed consent and assent forms.

Baseline data collection Parents and teachers will complete baseline questionnaires via online form.

Randomization After baseline questionnaires for a child participant are completed by parent and teacher, the child's family will be randomly assigned to the Mightier Now study cohort or the Mightier Later study cohort.

Before enrollment starts, a randomization list 60 subjects long will be created. Participants will be assigned to groups per this list, in the same order in which participants enroll in the study.

Intervention Families in the Mightier Now cohort will receive a Mightier shipment via UPS and will be directed to encourage child participants to play Mightier in their homes on an ad lib basis for eight weeks. Families in the Mightier Later cohort will be advised that their Mightier shipment will arrive after Week 8 questionnaires have been completed by a parent and teacher of the child participant.

Study check-ins Research staff will check in with families at weeks 0, 2, 4, and 6 of the study.

Study check-ins will consist of:

An email from research staff acknowledging child cumulative Mightier play minutes and encouraging ongoing play, Mightier gameplay engagement support, and links for scheduling study phone calls or zoom calls, at the discretion and preference of study participants.

Safety monitoring Participant safety will be assessed at study visits. Adverse events will be monitored and recorded. Concerns about participant safety will be reviewed by a clinician-on-call, a licensed clinical social worker, who will aid with referrals to local authorities as necessary.

Follow-up data collection Parents and teachers will complete follow-up questionnaires via online form as close as possible to 8 weeks after start of play.

Duration of treatment:

8 weeks of use ad-libitum. Parents in the Mightier Now study cohort will be encouraged to have their children play Mightier games at least 3 times a week / at least 45 minutes per week of Mightier play for the 8 week duration.

Parents in the Mightier Later study cohort will be reminded that they are in a "wait list" cohort, and that their Mightier shipment will arrive after parents and teachers complete the baseline and follow-up questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-11 at the time of screening
* Attending school outside of the home and not planning to change schools or classrooms during the 8-week study period

Exclusion Criteria:

* Prior Mightier use
* Out-of-home School Teacher unable to complete baseline and follow-up questionnaires
* Planned medication changes during the 8-week study period
* Parents encouraged to self-exclude if their children have severe skin sensitivities
* Parents encouraged to self-exclude if their children are pre-readers

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 43 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in in-school problem behaviors from baseline to follow-up | Baseline and Week 8
  Child Behavior Checklist- Teacher Report Form (CBCL-TRF): The CBCL-TRF (Achenbach & Rescorla, 2001) assesses child adaptive behaviors and problem behaviors. There are 112 items that assess problem behaviors and 16 items that assess academic performance and adaptive behavior. School teachers of child participants will complete the CBCL-TRF at baseline and Week 8.
Change in in-home problem behaviors from baseline to follow-up | Baseline and Week 8
  Child Behavior Checklist (CBCL/6-18): The CBCL/6-18 (Achenbach & Rescorla, 2001) assesses child adaptive behaviors and problem behaviors. There are 112 items that assess problem behaviors and 20 items that assess adaptive behavior. Response format for problem behaviors is from 0 ("not true") to 2 ("very true"). Parent participants will complete the CBCL/6-18 at baseline and follow-up.
Change in irritable mood from baseline to follow-up | Baseline and Week 8
  Affective Reactivity Index- Parent Report (ARI-P): The ARI is a 7-item scale that consists of 6 symptom items and 1 impairment item. The scale was designed to determine irritable mood rather than behavioral consequences such as hostility and acts of aggression (Stringaris et al., 2012). The individual items are scored 0,1, 2, and only the first six items are summed to form the total score, with a minimum score of 0 and a maximum score of 18, and higher scores indicating greater severity of irritability symptoms. The seventh item is an impairment item and it is analysed separately, with a minimum score of 0 and a maximum score of 3, and higher scores indicating greater irritability symptom severity. Parent participants will complete the ARI-P at baseline and Week 8.
Overall emotional regulation improvement as reported by teacher | Week 8
  Clinical Global Impressions Scale Improvement Question (CGI-I): The CGI is a self-report question that asks the respondent if they have noticed any overall improvements in the child's emotion regulation, with response options ranging from (1) very much improved to (7) very much worse. The Teacher CGI-I has not been scientifically validated for use in research studies. Teachers of child participants will complete the CGI-I at follow-up.
Overall emotional regulation improvement as reported by parent | Week 8
  Clinical Global Impressions Scale Improvement Question (CGI-I): The CGI is a self-report question that asks the respondent if they have noticed any overall improvements in the child's emotion regulation, with response options ranging from (1) very much improved to (7) very much worse. The Parent CGI-I has not been scientifically validated for use in research studies. Parents of child participants will complete the CGI-I at follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuromotion Labs, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ducharme P, Kahn J, Vaudreuil C, Gusman M, Waber D, Ross A, Rotenberg A, Rober A, Kimball K, Peechatka AL, Gonzalez-Heydrich J. A "Proof of Concept" Randomized Controlled Trial of a Video Game Requiring Emotional Regulation to Augment Anger Control Training. Front Psychiatry. 2021 Sep 1;12:591906. doi: 10.3389/fpsyt.2021.591906. eCollection 2021. PMID 34539455
- [Background] Achenbach, T. M., & Rescorla, L. A. (2001). Manual for the ASEBA School-Age Forms & Profiles. Burlington, VT: University of Vermont, Research Center for Children, Youth, & Families.
- [Background] Stringaris A, Goodman R, Ferdinando S, Razdan V, Muhrer E, Leibenluft E, Brotman MA. The Affective Reactivity Index: a concise irritability scale for clinical and research settings. J Child Psychol Psychiatry. 2012 Nov;53(11):1109-17. doi: 10.1111/j.1469-7610.2012.02561.x. Epub 2012 May 10. PMID 22574736
- [Background] Guy, WBRR (1976). CGI. Clinical global impressions. ECDEU assessment manual for psychopharmacology.